CLINICAL TRIAL: NCT05221268
Title: Effect of Repeated Downhill Walking Bouts on Ankle Isokinetic Parameters in Children With Obesity
Brief Title: Effect of Downhill Training on Ankle Joint
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taif University (Other)
Responsible Party: Principal Investigator, Hatem Allam, Assitant prof., Taif University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 646
Record Dates: First submitted 2021-12-20; First posted 2022-02-02 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- downhill (Experimental): Received downhill walking training.
  Interventions: Other: Downhill exercise
- Level -walking (Experimental): Received level walking training.
  Interventions: Other: Level walking exercise

INTERVENTIONS:
Other: Level walking exercise — treadmill exercise with 0 inclination
  Arms: Level -walking
Other: Downhill exercise — treadmill exercise with -20 inclination
  Arms: downhill

SUMMARY:
Downhill training help to improve musculoskeletal condition. Applying downhill training could help obese children by improving their muscular strength.

DETAILED DESCRIPTION:
the current study aimed to find the effect of downhill training on the ankle isokinetic parameters of obese children. There were two experimental groups, the first received level walking while the second received downhill training. The ankle isokinetic parameters were assessed pre and post-intervention for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index percentile 95% or more
* age ranged from 8-12 year
* student in one of Taif's elementary schools

Exclusion Criteria:

* suffering from any musculoskeletal problem or chronic disease.
* engaged in regular sports activities during the last 6 months

Ages: 8 Years to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2021-12-05 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Isokinetic eccentric plantarflexion tourque | 6 weeks
  Eccentric plantarflexion normalized peak tourque N.M/kg
Isokimetic Concentric plantarflexion tourque | 6 weeks
  Concentric dorsiflexion normalized peak tourque N.M/kg
Isokinetic Eccentric dorsiflexion tourque | 6 weeks
  Eccentric dorsiflexion normalized peak tourque N.M/kg
Isokinetic Concentric dorsiflexion tourque | 6 weeks
  Concentrc dorsiflexion normalized peak tourque N.M/kg

CONTACTS AND LOCATIONS:
Locations (1):
- College of applied medical sciences, Ta'if, Mecca Region, Saudi Arabia